CLINICAL TRIAL: NCT04891562
Title: Rhythmic Interlimb Coordination in Children with Developmental Coordination Disorder Compared to Typical Developing Children: the Effect of Individual, Task and Environmental Constraints
Brief Title: Rhythmic Interlimb Coordination in Children with Developmental Coordination Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Eugene Rameckers, Principal Investigator, Hasselt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RIC-CHILD-001
Record Dates: First submitted 2021-05-13; First posted 2021-05-18 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Developmental Coordination Disorder
Keywords: Developmental Coordination Disorder; Interlimb coordination; Gait; Sensorimotor synchronization; Metronomes
MeSH Terms: conditions — Motor Skills Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- pDCD (hildren with (probably) Developmental Coordination Disorder) (Experimental): children with (probably) Developmental Coordination Disorder (pDCD)
  Interventions: Other: interlimb coordination of the lower limbs and synchronization
- TDC (Typically Developing Children) (Active Comparator): Typically Developing Children
  Interventions: Other: interlimb coordination of the lower limbs and synchronization

INTERVENTIONS:
Other: interlimb coordination of the lower limbs and synchronization — 4 sessions (2 descriptive sessions, 2 experimental sessions), each lasting around 60 minutes. The m-ABC2 test, The MBEMA-s, Kids BESTest, interlimb coordination and synchronization investigation (visit 3 and 4)

SUMMARY:
This study is a case-controlled observational study, involving children with Developmental Coordination Disorder (DCD) and typically developing children with an age from 8 up to 12 years old. The study aims to investigate interlimb coordination of the lower limbs and sensorimotor synchronization ability in children with DCD compared to age-matched typically developing children during gait and fundamental lower limb coordination task to 2 metronomes with different temporal structures. The study consists of a maximum of 4 sessions (2 descriptive sessions, 2 experimental sessions), each lasting around 60 minutes. Depending on the preferences of the child and parents, the sessions can be combined in 2 sessions of 2 hours. During the first descriptive session, the participant will perform the m-ABC2 test to assess gross and fine motor function. The MBEMA-s will be used to examine rhythm perception ability. During the second descriptive session, children will perform the Kids BESTest to examine postural control, and two cognitive tests (digit span, go-no/go test) to assess executive functioning. During the third visit (experimental session), interlimb coordination and synchronization will be investigated during three tasks with different dynamic balance demands (seated, walking and running) in three conditions: in silence, to beats in isochronous metronome (discrete structure), to beats in non-isochronous metronomes (sinusoidal structure). In the last experimental session, the tempi of the auditory metronomes will be set at higher and lower tempi than the preferred comfortable tempo of the child.

ELIGIBILITY:
Inclusion Criteria:

* are aged between 8-12 years
* have no medical conditions that could impede their motor abilities.
* Children with a diagnosis of DCD, consistent with the DSM-V (Blank et al., 2019), or total percentile score <P16 on the movement assessment battery for children edition 2 (m-ABC-2), will be included in the group of (probably) DCD.
* The m-ABC score total of typical developing children needs to be ≥P25 for inclusion

Exclusion Criteria:

• have other neurological, orthopaedical, cardiorespiratory or intellectual impairment that could affect their motor abilities (verified using a health questionnaire)

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-01-18 (Actual)

PRIMARY OUTCOMES:
Phase coordination index (PCI) | week 2
  PCI is a measurement of consistency and accuracy in generating a series of anti-phase left - right stepping phases. Detailed information is described in Plotnik et al. (2007). Shortly, phase represent the relative timing of contralateral heel strikes, determining the phase, and normalize the step time with respect to the stride time (Plotnik, Giladi, & Hausdorff, 2007). Ideal interlimb coordination for each step is 180°. The consistency of the phase generation is represented by the Coefficient of variation of the series of the relative timing of the stepping of one leg with respect to the gait cycle.A lower PCI%, closer to zero, indicates a better antiphase interlimb coordination pattern.
Phase coordination index (PCI) | week 3
  PCI is a measurement of consistency and accuracy in generating a series of anti-phase left - right stepping phases. Detailed information is described in Plotnik et al. (2007). Shortly, phase represent the relative timing of contralateral heel strikes, determining the phase, and normalize the step time with respect to the stride time (Plotnik, Giladi, & Hausdorff, 2007). Ideal interlimb coordination for each step is 180°. The consistency of the phase generation is represented by the Coefficient of variation of the series of the relative timing of the stepping of one leg with respect to the gait cycle.A lower PCI%, closer to zero, indicates a better antiphase interlimb coordination pattern.
Auditory motor coupling - Resultant Vector Length to quantify synchronization consistency | week 2
  Synchronization consistency of steps to the beats during walking and running; and of the knee flexion-extension movement to the beats during the seated task
  Resultant Vector Length to quantify synchronization consistency. If the distribution of the relative phase angles over time is consistent, it results in a high resultant vector length (maximum value 1). If the synchronization is not consistent, the resultant vector length will be low (minimum value 0)
Auditory motor coupling - Resultant Vector Length to quantify synchronization consistency | week 3
  Synchronization consistency of steps to the beats during walking and running; and of the knee flexion-extension movement to the beats during the seated task
  Resultant Vector Length to quantify synchronization consistency. If the distribution of the relative phase angles over time is consistent, it results in a high resultant vector length (maximum value 1). If the synchronization is not consistent, the resultant vector length will be low (minimum value 0)
Auditory motor coupling - Relative phase angle | week 2
  Synchronization accuracy of steps to the beats during walking and running; and of the knee flexion-extension movement to the beats during the seated task. Relative phase angle, asynchrony in time to quantify synchronization accuracy (in degrees and in milliseconds respectively)
Auditory motor coupling - Relative phase angle | week 3
  Synchronization accuracy of steps to the beats during walking and running; and of the knee flexion-extension movement to the beats during the seated task. Relative phase angle, asynchrony in time to quantify synchronization accuracy (in degrees and in milliseconds respectively)

SECONDARY OUTCOMES:
velocity (m/s) | week 2
  Spatiotemporal parameters during the walking and running tasks:
  Gait velocity (m/s): absolute values, variability (standard deviation) of spatiotemporal parameters and values normalized to leg length will be reported.
velocity (m/s) | week 3
  Spatiotemporal parameters during the walking and running tasks:
  Gait velocity (m/s): absolute values, variability (standard deviation) of spatiotemporal parameters and values normalized to leg length will be reported.
step width (cm) | week 2
  Spatiotemporal parameters during the walking and running tasks:
  step width: absolute values, variability (standard deviation) of spatiotemporal parameters and values normalized to leg length will be reported.
step width (cm) | week 3
  Spatiotemporal parameters during the walking and running tasks:
  step width: absolute values, variability (standard deviation) of spatiotemporal parameters and values normalized to leg length will be reported.
stride length (cm) | week 2
  Spatiotemporal parameters during the walking and running tasks are: stride length (cm): absolute values, variability (standard deviation) of spatiotemporal parameters and values normalized to leg length will be reported.
stride length (cm) | week 3
  Spatiotemporal parameters during the walking and running tasks are: stride length (cm): absolute values, variability (standard deviation) of spatiotemporal parameters and values normalized to leg length will be reported.
cadence (step/minute) | week 2
  Spatiotemporal parameters during the walking and running tasks cadence (step/minute): absolute values, variability (standard deviation) of spatiotemporal parameters and values normalized to leg length will be reported.
cadence (step/minute) | week 3
  Spatiotemporal parameters during the walking and running tasks cadence (step/minute): absolute values, variability (standard deviation) of spatiotemporal parameters and values normalized to leg length will be reported.
double support (%gait cycle) | week 2
  Spatiotemporal parameters during the walking and running tasks:
  double support. Absolute values, variability (standard deviation) of spatiotemporal parameters and values normalized to leg length will be reported.
double support (%gait cycle) | week 3
  Spatiotemporal parameters during the walking and running tasks:
  double support. Absolute values, variability (standard deviation) of spatiotemporal parameters and values normalized to leg length will be reported.
movement frequency | week 2
  Spatiotemporal parameters during the seated antiphase knee flexion- extension task: movement frequency. The movement frequency of the leg movement signifies the temporal movement parameter, expressed as the amount of movement cycles in one minute. One movement cycle is defined between two successive peak extension positions. The average movement frequency of each leg, per metronome condition, will be calculated.
movement frequency | week 3
  Spatiotemporal parameters during the seated antiphase knee flexion- extension task: movement frequency. The movement frequency of the leg movement signifies the temporal movement parameter, expressed as the amount of movement cycles in one minute. One movement cycle is defined between two successive peak extension positions. The average movement frequency of each leg, per metronome condition, will be calculated.
movement amplitude | week 2
  Spatiotemporal parameters during the seated antiphase knee flexion- extension task: movement amplitude. The movement amplitude of the leg movement signifies the spatial movement parameter, for each individual movement cycle. The average amplitude of the movement cycles per metronome condition, for each leg separately, will be calculated.
movement amplitude | week 3
  Spatiotemporal parameters during the seated antiphase knee flexion- extension task: movement amplitude. The movement amplitude of the leg movement signifies the spatial movement parameter, for each individual movement cycle. The average amplitude of the movement cycles per metronome condition, for each leg separately, will be calculated.
The m-ABC (second edition) | Baseline
  The m-ABC (second edition) is a test to assess gross (static and dynamic balance, aiming and catching) and fine motor functions (manual dexterity) in children aged between 3 and 16 years. The m-ABC-second edition is a norm referenced test. The raw score of each task will be converted to standard scores (mean standard score of 10, standard deviation of 3) and percentiles. A lower score indicates a lower motor functioning. A total test score percentile below percentile 16 is at risk for problems with motor functions.
Montreal Battery of Evaluation of Musical Abilities (MBEMA-s) | Baseline
  beat perception ability will be assessed using two components (rhythm and melody) of the short version of the Montreal Battery of Evaluation of Musical Abilities (MBEMA-s). A maximum score of 20 can be attained for each component (rhythm and melody). A higher score indicated a better beat perception ability.
Kids BESTest | week 1
  Balance Evaluation Systems test for children" (Kids BESTest) includes six domains: biomechanical constraints (maximum score 15) , stability limits and verticality (maximum score 21), transitions/anticipatory (maximum score 18), Reactive(maximum score 18) , sensory orientation (maximum score 15), and stability in gait(maximum score 21) .For each task, a score of 0 indicates severe, where a score of 3 indicates normal performance. A higher score (total maximum score of 108) indicates a higher balance control.
digit span | week 1
  The digit span (forwards and backwards will be used to describe working memory. Children will be asked to listen to the digit span, consisting of random digits ranging from 1 to 9, and repeat the digit span forwards or backwards. The maximum length of digits that can be obtained is 9 for the digit span forward and 8 for the digit span backward. A higher score indicates a better performance.
go-no/go test | week 1
  The Go-no/Go task paradigm was developed to assess behavioral inhibition in children with limited working memory demands. Two versions of the Go-no/go test will be performed, namely an auditory and a visual.For both the auditory and visual task, a maximum score of 60 correct responses can be obtained. A lower score (minimum 0 correct) indicates a worse performance.

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Rameckers, prof. dr., Principal Investigator — Hasselt University; Mieke Goetschalckx, drs., Study Chair — Hasselt University
Locations (1):
- Hasselt University, Hasselt, Belgium

IPD SHARING:
Plan to Share IPD: No